CLINICAL TRIAL: NCT06845618
Title: Mycobacterium Tuberculosis Complex Cell-free DNA (Mtb-cfDNA) for the Pharmacometric Assessment of Anti-tuberculosis Treatment: a Proof-of-concept Study
Brief Title: Blood Tuberculosis DNA Levels to Monitor Tuberculosis Treatment
Acronym: Mtb-Dynamic
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: MYC24003
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-02

CONDITIONS: Mycobacterium Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Extra-Pulmonary
Keywords: cfDNA
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Extrapulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological specimens will be collected, processed, stored and shipped in concordance with established standard operating procedures. Blood will be collected following best practice venepuncture technique. Blood samples will be transferred by vehicle to the main SMRU laboratory in a cool box within six hours.
  The leftover blood samples will be stored and may be used for future studies for up to 30 years. Anonymised samples may be shared with collaborators internationally for further analysis. Consent will be obtained from participants for sample storage and future use of specimen. Any proposed plans to use samples other than for those investigations detailed in this protocol will be submitted to the relevant ethics committees prior to any testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Assay development and validation: Twenty participants with a new diagnosis of tuberculosis will have venous blood collected prior to treatment initiation. Twenty participants without clinical evidence of tuberculosis infection will be recruited from the local community as a control during assay validation. This group of the study participants will be assessed at day zero only.
- Group 2: Longitudinal Assessment: In this group, tuberculosis participants (n= 120) will have longitudinal sampling performed from diagnosis to the end of treatment. This will establish the feasibility of dynamic Mtb-cfDNA measurements for the assessment of tuberculosis treatment response.

SUMMARY:
Tuberculosis (TB) is a leading infectious cause of death worldwide. Current strategies for monitoring TB treatment response are culture dependent and insensitive. New methods of assessing treatment response in vivo could inform new drug development and other treatment strategies. Cell-free DNA (cfDNA) - small circulating fragments of DNA - is widely used in maternofetal medicine and oncology for diagnosis and assessment of treatment response. This study aims to investigate whether pathogen derived Mycobacterium tuberculosis-specific cfDNA (Mtb-cfDNA) can be used to monitor TB treatment response.

This feasibility study will take place at Mae RaMat TB Center in Thailand and includes two study groups:

1. Assay Development and Validation
2. Longitudinal Assessment of Mtb-cfDNA levels

DETAILED DESCRIPTION:
This study is funded by the Wellcome Trust; grant reference number: 223099/Z/21/Z

ELIGIBILITY:
Inclusion Criteria:

Participants with a new diagnosis of tuberculosis

* Aged ≥ 18 years old
* Newly microbiologically confirmed (culture or nucleic acid amplification test) diagnosis of Mycobacterium tuberculosis (Mtb.) infection (of any site)
* Has not yet commenced antituberculosis therapy
* Able to understand study procedures and requirements and is able to give informed consent

For healthy volunteers:

* Aged ≥ 18 years old
* Healthy as judged by a responsible physician
* Able to understand study procedures and requirements and is able to give informed consent

Exclusion Criteria:

Participants with a new diagnosis of tuberculosis

* Exposure to antituberculosis treatment in the last 8 weeks (or Mycobacterium tuberculosis (Mtb.) active fluoroquinolone)
* Known history of underlying malignancy
* Pregnancy
* Transfusion dependent anaemia

For healthy volunteers:

* History of tuberculosis infection or latent tuberculosis infection
* Household, or other close contact, of a person living with tuberculosis disease
* Chest radiograph (CXR) changes suggestive of pulmonary tuberculosis
* Presence of symptoms which would otherwise indicate screening for tuberculosis (cough > 2 weeks duration, fever, weight loss, night sweats)
* Other major medical comorbidity
* Pregnancy
* Known malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Assay development and validation. In this group, sampling will be performed at tuberculosis diagnosis. Tuberculosis participants (n = 20) will have blood sampling performed at day 0. Healthy participants (n = 20) without clinical evidence of tuberculosis will have blood sampling performed at a single timepoint.
  Group 2: Longitudinal Assessment. In this group, tuberculosis participants (n= 120) will have longitudinal sampling performed from diagnosis to the end of treatment. This will help to establish the feasibility of dynamic Mtb-cfDNA measurements.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Mtb-cfDNA trajectories | Day 0 - 168 (or end of treatment)
  Rate of Mtb-cfDNA clearance derived from serial Mtb-cfDNA measurements
Percentage of participants completing sampling schedule | Day 0 - 168 (or end of treatment)

SECONDARY OUTCOMES:
Exploratory analysis is planned and will compare Mtb-cfDNA levels to clinical, microbiological and radiological features | Day 0 - 168 (or end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Seers, Dr, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit, Faculty of Tropical Medicine, Mahidol University.
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The data generated in this study belongs to the study group as a whole. The final database will be shared amongst the PI and key members of the research team.
  With participant's consent, clinical data and results from blood analyses stored in the database may be shared with researchers not directly involved in this study but only after the main paper has been published and in accordance with MORU guidelines on data sharing.
  The results of the study will be summarised in lay language, in both English and the language(s) commonly spoken at the study site, and disseminated to participants and the community.
  The Investigators will be involved in reviewing drafts of the manuscripts, abstracts, press releases and any other publications arising from the study. Authorship will be determined in accordance with the International Committee of Medical Journal Editors (ICMJE) guidelines and other contributors will be acknowledged.